CLINICAL TRIAL: NCT02221804
Title: The Effect of Two Weeks of Voluntary Reduced Physical Activity in COPD - A Novel Methodology for Anabolic Drug Development
Brief Title: The Effect of Two Weeks of Voluntary Reduced Physical Activity in Chronic Obstructive Pulmonary Disease (COPD)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2014LF002B
Record Dates: First submitted 2014-08-18; First posted 2014-08-20 (Estimated); Last update posted 2014-08-22 (Estimated); Status verified 2014-08

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD); Muscle Atrophy
Keywords: Physical Inactivity; Skeletal Muscle; Cachexia
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Muscular Atrophy; Sedentary Behavior; Cachexia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- COPD - reduced activity levels (Experimental): COPD patients who have voluntarily decreased their daily physical activity levels to no more than 1500 steps/day for 14 days.
  Interventions: Behavioral: 14 days of voluntary step count reduction to no more than 1500 steps/day.
- Healthy - reduced activity levels (Experimental): Healthy age-matched controls who have voluntarily decreased their daily physical activity levels to no more than 1500 steps/day for 14 days.
  Interventions: Behavioral: 14 days of voluntary step count reduction to no more than 1500 steps/day.
- COPD - unchanged activity levels (No Intervention)

INTERVENTIONS:
Behavioral: 14 days of voluntary step count reduction to no more than 1500 steps/day.
  Arms: COPD - reduced activity levels; Healthy - reduced activity levels

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is the most common pulmonary disease, responsible for considerable morbidity and mortality and is the third leading cause of death worldwide. As well as its consequences in the lungs, COPD is well recognized to be associated with a range of important systemic consequences and co-morbidities. Interestingly, skeletal muscle dysfunction is noted in both early and advanced disease, suggesting its origins may not be wholly pulmonary.

Treatment strategies targeting lung function are, unfortunately, of limited value. Given the burden of disease, it is becoming increasingly important that investigative and therapeutic work now focuses on other systemic characteristics and sequelae which define the disease phenotype.

This is a randomized controlled trial of the effect of 14 days of voluntary reduced activity on muscle mass, muscle strength, body composition, and atrophy signalling in patients with COPD and age-matched controls.

The primary hypothesis upon which this study is based is that a short reduction in ambulation will induce a transient reduction in quadriceps muscle mass, quadriceps strength and physical performance in patients with COPD compared to matched COPD patients whose mobility has not been restricted.

The secondary hypothesis is that the magnitude of the above changes will be greater in physically inactive COPD patients compared to physically inactive age-matched controls.

The overall aim of this research is to use an in vivo human model of 14 days of voluntary reduced physical activity to test the above hypotheses. If the model proves feasible, this will allow for earlier proof of concept studies of novel therapeutic agents.

DETAILED DESCRIPTION:
This is a non-commercial randomized controlled trial. 15 patients with COPD and 15 age-matched controls will voluntarily reduce their daily step-count to no more than 1500 steps/day, from a baseline of > 3500 steps/day.

Before and after 14 days of reduced daily step-count, these 30 participants will undergo measures of appendicular mass, quadriceps strength, exercise tolerance and blood and urinary biomarkers. Quadriceps muscle biopsies will also be taken before and after the 14-day intervention.

15 patients with COPD will be studied 14 days apart but will not undergo the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking adult patients with COPD (GOLD stage II-IV)
* Non-smoking, healthy, age-matched controls
* Baseline step count > 3500 steps/day
* Baseline 6 minute walk distance > 140m

Exclusion Criteria:

* Inability to provide written, informed consent
* Significant co-morbidity limiting exercise tolerance
* Within 1 month of acute exacerbation of COPD
* Within 1 month of pulmonary rehabilitation
* History of venous thrombo-embolism or known increased risk of thrombotic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2014-05; Primary Completion 2016-04 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Quadriceps muscle mass as measured by dual-energy x-ray absorptiometry (DEXA) after two weeks of voluntary reduced physical activity. | Change from baseline in quadriceps muscle mass at 14 days.
  Dual-energy X-ray absorptiometry (DEXA) scanning will be used to assess body composition.
  Two X-ray beams with different energy levels are used during this technique. It is a widely used scanning modality and is entirely painless. The radiation received by the patient during the scan is less than that of an airline flight from California to New York and back.
  Specifically, appendicular lean composition will be measured (g).

SECONDARY OUTCOMES:
Quadriceps strength determined as maximal voluntary contraction force (QMVC) and the force elicited by unpotentiated supramaximal stimulation of the femoral nerve (TwQ). | Before and after the 14 day intervention
  Subjects sit on a specially designed chair keeping the knee flexed at 90 degrees over the end. Force is measured via an inextensible strap placed around the ankle and connected to a strain gauge. Subjects are asked to extend their knee maximally against the strap with visual feedback and verbal encouragement from the investigator, until no further increased in QMVC occurs.
  QMVC is reported in kg and is the highest single value obtained.
  In addition, the strength and endurance of the quadriceps will be measured using magnetic femoral nerve stimulation (TwQ). This is used to determine muscle strength in a non-volitional manner. The nerve to be studied is depolarised by the application of a rapidly changing magnetic field produced by a coil positioned on the overlying skin surface. The magnetic field is relatively unimpeded by skin, fat and bone, and thus has the ability to stimulate deep nerves easily and with little discomfort.
Rectus Femoris Cross Sectional Area determined by Quadriceps Ultrasound (RFCSA US) | Before and after the 14 day intervention
  An ultrasound (US) scan is a painless test that uses sound waves to create images of organs and structures. We will use it to assess the thickness of the thigh muscles.
  The patient rests in a reclined position for this test, and a lubricating jelly is applied to the thigh. The US probe is moved over the thigh area to produce a picture of the size of the thigh muscle. The leg to be scanned will be the same leg used for QMVC.
  The units of measure for the RFCSA are cm2.
6 minute walk distance (6MWD) | Before and after the 14 day intervention
  The 6MWD is a practical and simple test that measures the distance that a subject can walk quickly on a flat, hard surface in a period of 6 minutes. This will be performed by appropriately trained study site personnel.
  The outcome of the 6MWD will the walking distance covered in meters. The test will be performed according to the ATS Guidelines, in a standardized manner.
Short Physical Performance Battery (SPPB) | Before and after the 14 day intervention
  The SPPB is a brief performance test used to assess how well a subject can perform simple movements that represent the foundation of daily activities. The components that are assessed are 1) a Standing Balance Test, 2) a Four Meter Gait Speed and 3) a Sit to Stand Test. This collection of tests is routinely used in gerontology.
  It is scored out of a total of 12 points (4 for each of the 3 parameters aforementioned).
Blood and urinary biomarkers | Before and after the 14 day intervention
  Serum and plasma aliquots will be prepared from the blood samples for mediator analysis. Analysis will include full blood count, urea and electrolytes, d-dimers, and markers of systemic inflammation (C-reactive protein & fibrinogen). Each donation of blood will not exceed 50mL per study visit.
  Urine samples will be collected and frozen. These will be available for testing potentially relevant biomarkers which may come under investigation within our group.
Atrophy signalling determined from muscle biopsies | Before and after the 14 day intervention
  Muscle biopsies will be taken from the leg quadriceps muscle. These will be assessed for the presence of atrophy and hypertrophy signalling changes. The exact signalling panel will be determined from the most current literature review but is likely to include atrophic markers including myostatin, atrogin and MURF-1, hypertrophic markers including GSK3b, p70S6K and 4E-BP1, together with related microRNAs currently under investigation in our group.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Polkey, FRCP PhD, Principal Investigator — Royal Brompton & Harefield NHS Foundation Trust
Locations (1):
- Royal Brompton & Harefield NHS Foundation Trust, London, United Kingdom